CLINICAL TRIAL: NCT06981260
Title: The Role of Sound in Enhancing or Disabling the Placebo Effect of a Deactivated Transcutaneous Electrical Nerve Stimulator (TENS) Device on Hypoalgesia in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of Health and Resilience (Other)
Collaborators: Aegean College, Athens, Greece (Unknown); Coventry University, United Kingdom (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SOUNDPLACEBO-2016-001
Record Dates: First submitted 2025-05-07; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: A healthy volunteer pilot study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and assessor blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Placebo with sound (Experimental): Deactivated transcutaneous electrical nerve stimulation (TENS) with beeping sound (15-second interval)
  Interventions: Procedure: Group A Deactivated TENS with beeping sound (15-second interval)
- Group B: Placebo with no sound (Experimental): Group B: Deactivated transcutaneous electrical nerve stimulation (TENS) without sound
  Interventions: Procedure: Group B

INTERVENTIONS:
Procedure: Group A Deactivated TENS with beeping sound (15-second interval) — Deactivated TENS with beeping sound (15-second interval)
  Arms: Group A: Placebo with sound
Procedure: Group B — Deactivated TENS without sound
  Arms: Group B: Placebo with no sound

SUMMARY:
Placebo responses are now recognized for their clinical and physiological significance. Non-pharmacological cues such as sound may enhance or induce these responses. This trial aims to assess the effect of sound on the placebo-induced hypoalgesia elicited by a deactivated TENS device in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* No history of TENS use

Exclusion Criteria:

* Current medication use
* Orthopedic, neurological, or systemic conditions
* Pregnancy (current and planned)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2016-06-14 (Actual); Study Completion 2016-06-14 (Actual)

PRIMARY OUTCOMES:
Change in pain pressure threshold (PPT) at L2 (lumbar spine) from baseline to post-intervention. | From Baseliine to 5 minutes
  Change in pain pressure threshold (PPT) at L2 (2nd lumbar vertebra) from baseline to post-intervention. Measured using pressure algometer (Wagner Force Dial FDK/FDN Series).

SECONDARY OUTCOMES:
Effect of gender on placebo response | From Baseliine to 5 minutes
  Effect of gender on placebo response (ANOVA analysis on post-treatment PPT)

IPD SHARING:
Plan to Share IPD: No